CLINICAL TRIAL: NCT02143557
Title: The Effectiveness of Low Fat Breast Milk for the Treatment of Chylothorax in Infants Following Cardiothoracic Surgery: A Pilot Study
Brief Title: Dietary Treatment of Infants With Chylothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Labatt Family Heart Centre (Other); Trainee award through Ontario Student Opportunity Trust Fund - The Hospital for Sick Children Foundation Scholarship (Unknown)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000011037; 1000037303 (Other: The Hospital for Sick Children Research Ethics Board)
Record Dates: First submitted 2014-05-12; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Chylothorax
Keywords: breast milk; infants; chylothorax; cardiac surgery; modified breast milk
MeSH Terms: conditions — Chylothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fat-Modified Breast Milk (Experimental): Infants in this arm of the study were fed their own mother's breast milk where the fat layer was removed by centrifugation. Prior to feeding, extra energy and nutrients were added to the defatted breast milk.
  Interventions: Other: Fat-Modified Breast Milk
- MCT-formula group (Active Comparator): Infants in this arm of the study were fed a MCT-containing medical food which is the current standard of care.
  Interventions: Other: MCT formula

INTERVENTIONS:
Other: Fat-Modified Breast Milk
  Arms: Fat-Modified Breast Milk
Other: MCT formula
  Arms: MCT-formula group

SUMMARY:
Chylothorax occurs in ~3 to 5 % of infants undergoing cardiac surgery. Standard treatment requires discontinuation of breast milk feeding, due to the abundance of long chain triglycerides, and transition to a medium chain triglyceride (MCT) based formula. Objective: To determine the effectiveness of fat-modified breast milk (MBM) for the treatment of chylothorax compared with MCT-formula. Hypothesis: The investigators primary hypothesis was that infants fed MBM would have more chyle drainage in the first 5 days after diagnosis compared to infants fed an MCT based formula which is the current standard of care. Design: Infants with chylothorax were eligible. Treatment infants (n=8) received mother's own milk that had been modified by removing the fat layer via centrifugation and adding MCT and nutrients to provide 67 kcal/mL and 11 g/100 mL protein (MBM group). Control infants (n=8) received an MCT-formula (MCT group). The feeding intervention was a minimum of 6 weeks after chest tube removal per The Hospital for Sick Children standard chylothorax treatment protocol. Outcome measures collected included chyle drainage from chest tubes, weight, length and head circumference measurements and estimated energy and nutrient intake.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 12 months of age who were diagnosed with chylothorax.
* Infants included in the intervention group (MBM) needed to have received >80% of their enteral feeds as breast milk prior to surgery.
* Infants included in the control group (MCT-formula) needed to have received <80% of their enteral feeds as breast milk prior to surgery.

Exclusion Criteria:

* Subjects were excluded if their diagnosis made it unlikely that they would be able to follow the hospital's standard 6 week protocol for treatment of chylothorax
* Were receiving only parenteral nutrition at the time of diagnosis of chylothorax
* Primary caregiver of the baby did not have good comprehension of English.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Chyle Drainage from Chest Tubes | 6 weeks of chylothorax treatment
  This outcome includes measurement of chyle drainage from chest tubes in the first 5 days after diagnosis of chylothorax and the number of days of chest tube drainage.

SECONDARY OUTCOMES:
Growth | 6 weeks of the chylothorax treatment
  Infant weight, length and head circumference measurements were determined at study initiation and at the first post-discharge follow-up visit (within one-week of discharge) and again at the end of chylothorax treatment.

OTHER OUTCOMES:
Estimated Nutrient Intakes | 6 weeks of chylothorax treatment
  Average daily energy, protein and other nutrient intakes were calculated using milk volumes consumed (recorded in the medical record [in-hospital] or 3 day consecutive food records [after discharge]), analyzed breast milk fat composition values, milk nutrient values from the literature, product monographs and Food Processor SQL Ed v. 10.2 (ESHA Research).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, PhD RD, Principal Investigator — The Hospital for Sick Children; Sarah Kocel, MSc RD, Principal Investigator — The Hospital for Sick Children; Jennifer Russell, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada